CLINICAL TRIAL: NCT04317742
Title: eHealth Insomnia Intervention for Adult Survivors of Childhood Cancer: A Randomized Clinical Trial
Brief Title: eHealth Insomnia Intervention for Adult Survivors of Childhood Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SLEEPWELL; 1R01CA239689 (NIH)
Record Dates: First submitted 2020-02-18; First posted 2020-03-23 (Actual); Results first posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Childhood Cancer; Insomnia; Neurocognitive Impairment; Survivorship; Late Effect; Sleep
MeSH Terms: conditions — Neoplasms; Sleep Initiation and Maintenance Disorders | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sleep Healthy Using the Internet (SHUTi) Intervention Group (Active Comparator): Participants access and complete the SHUTi program for 9 weeks.
  Interventions: Device: Sleep Healthy Using the Internet (SHUTi) Intervention Group
- Online Patient Education (PE) Control Group (Active Comparator): Participants access and review online patient education for 9 weeks.
  Interventions: Device: Online Patient Education (PE) Control Group

INTERVENTIONS:
Device: Sleep Healthy Using the Internet (SHUTi) Intervention Group — SHUTi is a fully automated, interactive and tailored web-based program that incorporates the primary tenets of face-to-face CBT-I, including sleep restriction, stimulus control, cognitive restructuring, sleep hygiene, and relapse prevention. Intervention content is presented in six "Cores," metered out over time.
  Arms: Sleep Healthy Using the Internet (SHUTi) Intervention Group
Device: Online Patient Education (PE) Control Group — The online PE program provides static information about: insomnia symptoms; the impact, prevalence, and causes of insomnia; when to see a doctor; and basic lifestyle, environmental, and behavioral strategies to improve sleep.
  Arms: Online Patient Education (PE) Control Group

SUMMARY:
There is evidence that survivors of childhood cancer have a high prevalence of poor sleep, including symptoms of insomnia. Insomnia is highly comorbid and has been associated with impaired cognitive performance, a range of psychiatric disorders, cardiovascular disease, and reduced quality of life. However, we still lack knowledge about the direct impact of available internet-based insomnia treatment programs for survivors of childhood cancer experiencing insomnia, in addition to how improving insomnia symptoms impacts neurocognitive function and late health morbidities in this population. Therefore, in this study, we will utilize the resources available in the Childhood Cancer Survivor Study (CCSS) to use an accepted, established, efficacious internet-delivered CBTi insomnia treatment program and evaluate the efficacy of this program in adult survivors of childhood cancer. Positive results from this study and our use of an internet-based intervention are likely generalizable and be scalable to the large and geographically diverse population of childhood cancer survivors with chronic health conditions.

Primary Objective

To examine the efficacy of an eHealth intervention for improving symptoms of insomnia among adult survivors of childhood cancer.

Secondary Objectives

To examine the impact of an eHealth intervention for insomnia on the clinical severity of insomnia symptoms in adult survivors of childhood cancer.

To determine whether treatment of insomnia symptoms will improve neurocognitive function in adult survivors of childhood cancer with both insomnia and neurocognitive impairment.

To explore the mediating effects of improved neurocognitive function, emotional distress, and cardiovascular health on the association between insomnia symptoms and quality of life.

DETAILED DESCRIPTION:
Participants with clinically significant insomnia and neurocognitive impairment are eligible for the current study. Participants will complete a 9-week internet-based insomnia treatment program (SHUTi) or receive sleep education, depending on randomized group assignment. Participants will complete home-based assessments at 3 time points (baseline, post-intervention, 6 months). These assessments will include online questionnaires measuring insomnia symptoms, neurocognitive problems, fatigue, daytime sleepiness, and health related quality of life. In addition, at each time point participants will be asked to wear an activity monitor for one week to measure physical activity and sleep patterns. Each assessment time point will also include assessment of cardiovascular biomarkers (dried blood spot cards) and neurocognitive function (CNS Vital Signs).

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in CCSS
* Between the ages of 18 and 65 years old
* Meeting at least one of the following three insomnia criteria:
* Clinically significant insomnia (i.e. score ≥8 on the Insomnia Severity Index)
* Delayed sleep onset latency (SOL) (i.e. cannot get to sleep within 30 minutes, three or more times a week)
* Excessive wake after sleep onset (WASO) (i.e. nighttime awakenings lasting a total of at least 30 minutes, three or more times per week)
* Neurocognitive impairment (i.e. score >84th %ile of sibling normative data in at least one domain on the CCSS-NCQ)
* Regular access to the internet (at least 2-3 days per week)
* Ability to read and speak English
* Access to a desktop computer or a laptop
* Access to a smart phone (android or iPhone), tablet or iPad with Bluetooth Low Energy BLE 4.2 or higher

Exclusion Criteria:

* History of a brain tumor
* An irregular schedule that would prevent adoption of intervention strategies (i.e. work schedule resulting in usual bedtime earlier than 8 PM or later than 2 AM or arising time earlier than 4 AM or later than 10 AM)
* Currently pregnant or breast feeding
* Behavioral treatment for insomnia in the past 12 months
* Diagnosis of schizophrenia or a psychotic disorder
* Alcohol or drug abuse in past year
* Other concurrent sleep disorders, including narcolepsy, obstructive/central sleep apnea, or restless leg syndrome
* Current treatment or intervention for cognitive impairment (i.e. stimulant medication, transcranial direct current stimulation)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1554 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tara Brinkman, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1554 participants were screened and enrolled between December 2020 and February 2024. Of these, 989 were ineligible, 9 withdrew and 15 were lost to follow-up prior to randomization. 541 participants were randomized.
Pre-assignment Details: The remaining 541 participants were randomized to complete the SHUTi intervention program or to review the online patient education materials for 9 weeks. Participants were randomized using a permuted-block method with random block sizes, stratified on sex (male/female), age (<40/>40), and cranial radiation therapy (yes/no).
Period: Overall Study
Arm/Group | Sleep Healthy Using the Internet (SHUTi) Intervention Group | Online Patient Education (PE) Control Group
Started (Participants enrolled and randomized to intervention arms.) | 273 | 268
Completed (Participants who completed baseline and post-intervention assessment.) | 169 | 184
Not Completed | 104 | 84
Not completed — Lost to Follow-up | 57 | 59
Not completed — Pregnancy | 1 | 1
Not completed — Withdrawal by Subject | 46 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sleep Healthy Using the Internet (SHUTi) Intervention Group | Online Patient Education (PE) Control Group | Total
Number analyzed (Participants) | 273 | 268 | 541
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.6 (8.7) | 44.8 (8.7) | 44.7 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197 | 198 | 395
  Male | 76 | 70 | 146
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 232 | 226 | 458
  Black, non-Hispanic | 10 | 7 | 17
  Hispanic | 19 | 18 | 37
  Other races, non-Hispanic | 10 | 16 | 26
  Unknown | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 273 | 268 | 541

OUTCOME MEASURES:

1. Primary Outcome: Change in Insomnia Severity Index (ISI) Scores From Baseline to Post-Intervention (Approximately 10 Weeks After Baseline)
Description: This is a 7-item, Likert scale, self-report questionnaire assessing perception of sleep and consequences of insomnia. The scores range from 0 to 28 with higher values indicating increasing symptom burden. Changes in scores on a scale from baseline to post-intervention are reported.
Time Frame: Baseline and Post-Intervention (approximately 10 weeks after Baseline)]
Population: Analysis based on intent to treat. Include participants who were randomized and completed both the baseline and 10-week post-intervention assessments.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sleep Healthy Using the Internet (SHUTi) Intervention Group | Online Patient Education (PE) Control Group
Number analyzed (Participants) | 169 | 184
Score on a scale | -6.30 (5.04) | -3.91 (4.62)

2. Secondary Outcome: Change in Childhood Cancer Survivor Study-Neurocognitive Questionnaire (CCSS-NCQ) Scores From Baseline to Post-Intervention (Approximately 10 Weeks After Baseline)
Description: The CCSS-NCQ was developed specifically to address neurocognitive concerns of adult survivors of childhood cancer and includes assessment of problems with memory, task efficiency, organization, and emotional regulation. The domains of memory, task efficiency, and emotional regulation are used in this study. Z-scores are calculated using sibling normative data (Mean=1, SD=0) with higher scores indicating worse problems. Changes in z-scores from baseline to post-intervention are reported.
Time Frame: Baseline and Post-Intervention (approximately 10 weeks after Baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sleep Healthy Using the Internet (SHUTi) Intervention Group | Online Patient Education (PE) Control Group
Number analyzed (Participants) | 169 | 184
Z-score
  Task efficiency | -0.70 (1.00) | -0.41 (0.92)
  Memory | -0.65 (1.01) | -0.36 (0.87)
  Emotional regulation | -0.66 (0.90) | -0.43 (0.81)

3. Secondary Outcome: Change in CNS Vitals Signs Scores From Baseline to Post-Intervention (Approximately 10 Weeks After Baseline)
Description: This is a computerized assessment that measures 3 domains of cognitive function; Executive Function, Processing Speed and Memory. Age, sex, and race specific Standard Scores (M=100, SD=15) are calculated. Higher scores indicate better functioning. Changes in standard scores from baseline to post-intervention are reported.
Time Frame: Baseline and Post-Intervention (approximately 10 weeks after Baseline)]
Population: Analysis based on intent to treat. Include participants who randomized and completed both the baseline and 10-week post-intervention assessments. Participants with missing or invalid CNS Vital Signs assessment in each domain (Executive function, n = 54; Memory, n = 48; Processing Speed, n=36) were removed.
Measure: Mean (Standard Deviation); unit: Standard score
Arm/Group | Sleep Healthy Using the Internet (SHUTi) Intervention Group | Online Patient Education (PE) Control Group
Number analyzed (Participants) | 169 | 184
Standard score
  Executive function | 1.9 (13.0) | 3.5 (11.8)
  Memory | 2.6 (15.7) | 0.1 (17.2)
  Processing speed | 3.9 (12.7) | 3.3 (11.9)

4. Secondary Outcome: Change in Patient Health Questionnaire (PHQ-8) Scores From Baseline to 6-Month Follow-Up (Approximately 6 Months After Baseline)
Description: This questionnaire measures symptoms of depression. Scores range from 0 to 24 with higher scores indicating more severe symptoms. Changes in scores on a scale from baseline to 6-month follow-up are reported.
Time Frame: Baseline and 6-Month Follow up (approximately 6 months after Baseline)
Population: Analysis based on intent to treat. Include participants who randomized and completed both the baseline and 6-month follow-up assessments.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sleep Healthy Using the Internet (SHUTi) Intervention Group | Online Patient Education (PE) Control Group
Number analyzed (Participants) | 137 | 168
Score on a scale | -2.7 (4.1) | -1.3 (4.3)

5. Secondary Outcome: Change in Generalized Anxiety Disorder-7 (GAD-7) Scores From Baseline to 6-Month Follow-up (Approximately 6 Months After Baseline)
Description: This questionnaire measures symptoms of anxiety with scores ranging from 0 to 21. Higher scores indicate greater symptoms of anxiety. Changes in scores on a scale from baseline to 6-month follow-up are reported.
Time Frame: Baseline and 6-Month Follow up (approximately 6 months after Baseline)
Population: Analysis based on intent to treat. Include participants who were randomized and completed both the baseline and 6-month follow-up assessment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sleep Healthy Using the Internet (SHUTi) Intervention Group | Online Patient Education (PE) Control Group
Number analyzed (Participants) | 137 | 168
Score on a scale | -2.3 (4.0) | -1.4 (4.6)

6. Secondary Outcome: Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health Questionnaire (HRQoL) Scores From Baseline to 6-Month Follow-up (Approximately 6 Months After Baseline)
Description: This questionnaire measures general health-related quality of life in the domains of physical and mental health. T-scores are calculated (M=50, SD=10) with higher scores indicated better quality of life. The PROMIS scoring tables were used for scoring. Changes in T-scores from baseline to 6-month follow-up are reported.
Time Frame: Baseline and 6-Month Follow up (approximately 6 months after Baseline)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Sleep Healthy Using the Internet (SHUTi) Intervention Group | Online Patient Education (PE) Control Group
Number analyzed (Participants) | 137 | 168
T-score
  Physical health | 2.5 (5.7) | 1.0 (5.3)
  Mental health | 2.6 (7.1) | 1.0 (6.3)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the overall study duration, from enrollment to 6-month follow-up, for each participant.
Description: Adverse events were self-reported by participants at any point during the study period.
Arm/Group | Sleep Healthy Using the Internet (SHUTi) Intervention Group | Online Patient Education (PE) Control Group
All-Cause Mortality (participants affected / at risk) | 0/273 | 0/268
Serious Adverse Events (participants affected / at risk) | 0/273 | 0/268
Other Adverse Events (participants affected / at risk) | 0/273 | 0/268

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/42/NCT04317742/Prot_SAP_000.pdf